CLINICAL TRIAL: NCT05935098
Title: A Phase 1a/1b Study Investigating the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Antitumor Activity of BGB-A3055, Alone and in Combination With Tislelizumab in Patients With Selected Advanced or Metastatic Solid Tumors
Brief Title: BGB-A3055 Alone and in Combination With Tislelizumab in Participants With Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BGB-A317-A3055-101; 2023-505322-34-00 (EU CTIS Number); CTR20241681 (Other: ChinaDrugTrials)
Record Dates: First submitted 2023-06-26; First posted 2023-07-07 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Advanced Solid Tumor; Metastatic Solid Tumor; Solid Tumor
Keywords: BGB-A3055; Tislelizumab; Advanced solid tumors; Safety monitoring; Monoclonal antibody; Preliminary antitumor activity; Metastatic cancer; Metastatic Solid Tumor; PD1; CCR8
MeSH Terms: conditions — Neoplasm Metastasis | interventions — tislelizumab; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase 1a Part A: Dose Escalation (BGB-A3055 Monotherapy) (Experimental): Different groups of participants will receive increasing doses of BGB-A3055 alone to determine the most appropriate dosage levels.
  Interventions: Drug: BGB-A3055
- Phase 1a Part B: Dose Escalation (BGB-A3055 + tislelizumab) (Experimental): Different groups of participants will receive increasing doses of BGB-A3055 in combination with tislelizumab to determine the most appropriate dosage levels.
  Interventions: Drug: BGB-A3055; Drug: Tislelizumab
- Phase 1b (Dose Expansion): (Experimental): Participants will receive the recommended dose for expansion (RDFE) of BGB-A3055 in combination with tislelizumab with or without chemotherapy to provide additional information on the safety, tolerability, and potential benefits of the recommended dose.
  Interventions: Drug: BGB-A3055; Drug: Tislelizumab; Drug: Chemotherapy

INTERVENTIONS:
Drug: BGB-A3055 — Administered intravenously
Drug: Tislelizumab — Administered intravenously
  Other Names: BGB-A317
  Arms: Phase 1a Part B: Dose Escalation (BGB-A3055 + tislelizumab); Phase 1b (Dose Expansion):
Drug: Chemotherapy — Administered in accordance with relevant local guidelines and/or prescribing information.
  Arms: Phase 1b (Dose Expansion):

SUMMARY:
This study aims to evaluate how safe and well-tolerated the treatment is, how the body processes it, how it works on the tumors, and whether it shows early signs of fighting cancer in people with certain advanced or metastatic solid tumors.

Key details of the study include:

* The study is expected to last about 36 months.
* Participants will receive treatment until they either no longer benefit from the treatment, experience side effects that are too severe, or choose to stop participating.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years on the day of signing the informed consent form (ICF) (or the legal age of consent in the jurisdiction in which the study is taking place, whichever is older).
2. All participants are also required to demonstrate an ECOG Performance Status score of ≤1 within 3 days before the first dose of study drug(s) and have adequate organ function.
3. Participants with histologically confirmed advanced or metastatic solid tumors associated with high CCR8 and who have previously received adequate available standard systemic therapy or for whom treatment is not available or not tolerated and who have not received any prior therapy targeting CCR8.
4. >=1 Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
5. Participants should be able to provide archival tumor tissue samples (as block or unstained slides) or fresh biopsy if there is no archival tissue at baseline. For selected cohorts, participants should be willing to provide post-treatment fresh biopsy at specified timepoints.
6. Females of childbearing potential and nonsterile males must be willing to use a highly effective method of birth control for the duration of the study, and for ≥ 120 days after the last dose of BGB-A3055 or tislelizumab (whichever is later), or up to 9 months after the last dose of chemotherapy, whichever is later. Females of childbearing potential must also have a negative urine or serum pregnancy test result ≤ 7 days before the first dose of study drug(s).

Exclusion Criteria:

1. Active leptomeningeal disease or uncontrolled, untreated brain metastasis.
2. Active autoimmune diseases or history of autoimmune diseases that may relapse
3. Any malignancy ≤ 3 years before the first dose of study drug(s) except for the specific cancer under investigation in this study and any locally recurring cancer that has been treated with curative intent (eg, resected basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the cervix or breast).
4. Participants with hepatitis B infection with HBV DNA ≥ 500 IU/mL (or ≥ 2500 copies/mL). Participants with active hepatitis C, and participants with HIV infection.

   Note: Participants with chronic hepatitis B infection or resolved hepatitis B infection (HBV DNA < 500 IU/mL or < 2500 copies/mL) and considered stable are eligible. Participants with a negative HCV antibody test result at screening or a positive HCV antibody test result followed by a negative HCV RNA test result at screening are eligible to participate. Participants with treated HIV infection may be included if certain criteria are met.
5. History of interstitial lung disease, noninfectious pneumonitis, or uncontrolled lung diseases including pulmonary fibrosis, or acute lung diseases.
6. Grade 3 immune-mediated adverse events on prior immune-oncology agent.
7. Cardiovascular risk factors, including but not limited to pulmonary embolism ≤ 28 days or history of acute myocardial infarction or heart failure ≤ 6 months before the first dose of study drug(s).
8. Uncontrolled diabetes.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 263 (Estimated)
Dates: Start 2023-08-21 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Phase 1a: Number of participants with adverse events (AEs) | Up to 2 Years
  Number of participants with treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) graded according to the National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0 and the American Society for Transplantation and Cellular Therapy [ASTCT] consensus grading system for cytokine release syndrome [CRS]), and including findings from laboratory assessments, electrocardiograms (ECGs), and physical examinations, and that meet protocol-defined dose-limiting toxicity (DLT) criteria.
Phase 1a: Maximum tolerated dose (MTD) or maximum administered dose (MAD) of BGB-A3055 | Up to 2 Years
  MTD is defined as the highest dose evaluated for which estimated toxicity rate is the closest to the target toxicity rate of 30%. MAD is defined as the highest dose administered.
Phase 1a: Recommended dose for expansion (RDFE) of BGB-A3055 alone or in combination with tislelizumab | Up to 2 Years
  The RDFEs of BGB-A3055, alone or in combination with tislelizumab will be determined based on biological effectiveness taking preclinical and clinical data, including safety, tolerability, pharmacokinetics (PK), pharmacodynamics, and antitumor activity, into consideration.
Phase 1b (Dose Expansion): Objective Response Rate (ORR) | Up to 2 Years
  ORR is defined as the percentage of participants who had complete response (CR) or partial response (PR) as assessed by the investigator per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.

SECONDARY OUTCOMES:
Phase 1a: ORR | Up to 2 Years
  ORR is defined as the percentage of participants who had complete response (CR) or partial response (PR) as determined from tumor assessments by the investigators per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
Time to Response (TTR) | Up to 2 Years
  Defined as the time from the date of the first administration of study drug(s) to the first determination of an objective response.as determined from tumor assessments by the investigators per RECIST v1.1.
Duration of Response (DOR) | Up to 2 Years
  Defined as the time from the first determination of an objective response to the time of first documentation of radiographic progression, as determined from tumor assessments by the investigators per RECIST v1.1, or death from any cause, whichever comes first.
Disease Control Rate (DCR) | Up to 2 Years
  Defined as the percentage of participants whose best overall response (BOR) is complete response, partial response, or stable disease as determined from tumor assessments by the investigators per RECIST v1.1.
Clinical Benefit Rate (CBR) | Up to 2 Years
  Defined as the percentage of participants whose best overall response (BOR) is complete response, partial response, or durable stable disease (stable disease for at least 24 weeks) as determined from tumor assessments by the investigators per RECIST v1.1.
Number of participants with anti-drug antibodies (ADAs) against BGB-A3055 | Up to 2 Years
Serum concentration of BGB-A3055 at specified time points | Up to 2 Years
Phase 1b: Progression-Free Survival (PFS) | Up to 2 Years
  Defined as the time from randomization to the first objectively documented disease progression, or death from any cause, whichever occurred first, as determined from tumor assessments by investigators per RECIST v1.1.
Phase 1b: Number of participants with adverse events (AEs) | Up to 2 Years
  Number of participants with TEAEs and SAEs graded according to the NCI-CTCAE version 5.0 and the ASTCT consensus grading system for CRS, and including findings from laboratory assessments, ECGs, and physical examinations.
Phase 1b: Association of CCR8 expression with clinical efficacy | Up to 2 Years
  Evaluated from participant-derived tumor tissue(s) obtained before and/or after treatment with BGB-A3055 in combination with tislelizumab with or without chemotherapy, and their association with clinical efficacy.
Phase 1b: Association of PD-L1 expression with clinical efficacy | Up to 2 Years
  Evaluated from participant-derived tumor tissue(s) obtained before and/or after treatment with BGB-A3055 in combination with tislelizumab with or without chemotherapy, and their association with clinical efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeiGene
Locations (26):
- United States (6):
  - Advent Health Cancer Institute, Orlando, Florida
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - John Theurer Cancer Center Hackensack University Medical Center, Hackensack, New Jersey
  - The University of Texas Md Anderson Cancer Center, Houston, Texas
  - Next Dallas, Irving, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- Australia (3):
  - Chris Obrien Lifehouse, Camperdown, New South Wales
  - Icon Cancer Centre South Brisbane, South Brisbane, Queensland
  - Linear Clinical Research, Nedlands, Western Australia
- China (9):
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Liaoning Cancer Hospital and Institute, Shenyang, Liaoning
  - Rui Jin Hospital Shanghai Jiao Tong University School of Medicinejiading Branch, Shanghai, Shanghai Municipality
  - Changzhi Peoples Hospital, Changzhi, Shanxi
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
- France (3):
  - Centre de Lutte Contre Le Cancer Institut Bergonie, Bordeaux
  - Institut Curie, Paris
  - Ico Site Rene Gauducheau, SaintHerblain
- South Korea (5):
  - Seoul National University Bundang Hospital, BundangGu SeongnamSi, Gyeonggi-do
  - Samsung Medical Center, GangnamGu, Seoul Teugbyeolsi
  - Severance Hospital Yonsei University Health System, SeodaemunGu, Seoul Teugbyeolsi
  - Seoul National University Hospital, Seoul, Seoul Teugbyeolsi
  - Asan Medical Center, SongpaGu, Seoul Teugbyeolsi

IPD SHARING:
Plan to Share IPD: Yes
BeiGene shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeiGene shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeiGene review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beigene.com/science/clinical-trials/